CLINICAL TRIAL: NCT01441037
Title: Male Hormones for Telomere Related Diseases
Brief Title: Danazol for Genetic Bone Marrow and Lung Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110209; 11-H-0209
Record Dates: First submitted 2011-09-24; First posted 2011-09-27 (Estimated); Results first posted 2018-07-11 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2017-12-18

CONDITIONS: Aplastic Anemia
Keywords: Aplastic Anemia; Androgen; Telomeres; Sex hormone; Pulmonary fibrosis; Liver cirrhosis
MeSH Terms: conditions — Anemia, Aplastic; Pulmonary Fibrosis; Liver Cirrhosis | interventions — Danazol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Danazol (Experimental): Single arm in which danazol is administered orally at 800 mg daily for 2 years.
  Interventions: Drug: Danazol

INTERVENTIONS:
Drug: Danazol — Danazol, 800 mg daily by mouth for 2 years

SUMMARY:
Background:

- Some people have bone marrow and lung disorders that are caused by genetic problems. These problems often involve damage to the ends of the chromosomes that pass down genes. One of these disorders is aplastic anemia. This is a disorder in which the bone marrow does not make enough blood cells. Currently, doctors use a male hormone-based drug called Danazol to improve bone marrow function and treat aplastic anemia. More information is needed on whether Danazol can help repair the damaged chromosomes that cause aplastic anemia and similar disorders that cause low blood cell counts or lung problems.

Objectives:

- To study the safety and effectiveness of Danazol for bone marrow and lung disorders caused by damaged genes.

Eligibility:

- Individuals at least 2 years of age who have low blood cell counts or lung fibrosis caused by damaged genes.

Design:

* Participants will be screened with a physical exam and medical history. Then they will have blood and urine tests, imaging studies, and a lung function test. They will also take a 6-minute walking test and have a bone marrow biopsy.
* Participants will receive Danazol to take twice a day for the duration of the study.
* Participants will have regular study visits at 6, 12, and 24 months, with blood tests, imaging studies, a lung function test, and a 6-minute walking test. A bone marrow sample will be collected at the 12-month visit.
* Participants will remain on the study for up to 2 years. Researchers will follow up with them for 2 years after the end of the study.

DETAILED DESCRIPTION:
Severe aplastic anemia (SAA) is a life-threatening bone marrow failure disorder characterized by pancytopenia and a hypocellular bone marrow. Telomeres were reported to be short in up to one-third of patients with SAA.Initially this occurrence was presumed to be secondary to hematopoietic stress. However, the discovery of loss-of-function mutations in genes of the telomerase complex (TERC, TERT) established a genetic etiology for telomere attrition in some patients with marrow failure who did not have the stigmata associated to an inherited bone marrow failure syndrome. These findings implicated telomerase dysfunction in failed hematopoiesis. In family members of probands with SAA, telomerase mutations have been observed which were associated to varying degrees of cytopenias, idiopathic pulmonary fibrosis (IPF) and/or cirrhosis.

Telomere length has been associated with human cancer. Telomere attrition has been implicated in a variety of solid organ malignancies including esophageal and colon adenocarcinoma. In a longitudinal population based study, shorter telomere length associated to a higher cancer mortality risk overtime. It is plausible that a shorter telomere length is not just a biomarker associated to development of cancer, but involved in its pathogenesis. Ample experimental data supports an important role of critically short telomere length in genomic instability. Furthermore, our laboratory data (unpublished) shows that similar chromosome instability occurs in bone marrow cells of mutant patients, confirming the experimental data. Thus, a common molecular mechanism appears to underlie risk for cancer and a range of clinical entities.

In vitro studies suggest that telomere length could, in theory, be modulated with sex hormones.15 Exposure of normal peripheral blood lymphocytes and human bone marrow derived CD34+ cells to androgens increased telomerase activity in vitro and androgens increased low baseline telomerase activity in individuals carrying a loss-of-function TERT mutation to normal levels. In retrospect, the beneficial effects of sex hormones on telomerase activity may be the mechanism by which SAA patients treated over 40 years ago with male hormones showed hematologic improvement in some cases.

In recent years we have seen patients referred to our clinic with varying degree of cytopenia(s) who had significant family history for cytopenia(s), IPF and/or cirrhosis. We have identified very short telomeres in these patients and in some mutations in TERC and TERT. We hypothesize that male hormone therapy might modulate telomere attrition in vivo and ameliorate progression or reverse the clinical consequences of accelerated telomere attrition. Therefore, we propose male hormone therapy in patients with cytopenia(s) and/or IPF who show evidence of telomere dysfunction by a short age adjusted telomere length associated to telomerase gene mutations. The primary biologic endpoint will be delay of telomere attrition over time compared to known rates of telomere erosion in normal individuals and in those who carry mutation in the telomerase genes. The main clinical endpoint will be tolerability of oral danazol over two years. Secondary endpoints will be improvement in blood counts and/or pulmonary function. The small sample size, lack of control groups, and variable clinical course among those with marrow failure and IPF, will not allow for definitive assessment of clinical benefit. Nevertheless, we believe this protocol will provide insight into the possible effects of androgen therapy on telomere attrition in humans and of possible clinical benefit in telomere related disorders, and serve as hypothesis generating for further larger controlled studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Short age-adjusted telomere length in the first percentile and/or a mutation in telomerase genes
  2. One or more of the following cytopenia(s).
* Anemia

  1. Symptomatic anemia with a hemoglobin < 9.5 g/dL or red cell transfusion requirements > 2 units/month for at least 2 months
  2. Reticulocyte count < 60,000 /microL
* Thrombocytopenia

  1. Platelet count < 30,000 /microL or < 50,000 /microL associated with bleeding
  2. Decreased megakaryocytic precursors in the bone marrow
* Neutropenia

  1. Absolute neutrophil count < 1,000 /microL

     OR

     3. Idiopathic pulmonary fibrosis diagnosed by either a lung biopsy of high resolution computed tomography scan of the chest according to guidelines from the American Thoracic Society and European Respiratory Society

     4. Age greater than or equal to 2 years

     5. Weight > 12 kg

     EXCLUSION CRITERIA:
     1. Moribund status or concurrent hepatic, renal, cardiac, neurologic, pulmonary, infectious, or metabolic disease of such severity that it would preclude the patient s ability to tolerate protocol therapy, or that death within 30 days is likely
     2. Potential subjects with cancer who are on active chemotherapeutic treatment
     3. Current pregnancy, or unwillingness to avoid pregnancy if of childbearing potential
     4. Not able to understand the investigational nature of the study or give informed consent or does not have a legally authorized representative or surrogate that can provide informed consent.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-07-19; Primary Completion 2016-11-14 (Actual); Study Completion 2016-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal S Young, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Young NS, Calado RT, Scheinberg P. Current concepts in the pathophysiology and treatment of aplastic anemia. Blood. 2006 Oct 15;108(8):2509-19. doi: 10.1182/blood-2006-03-010777. Epub 2006 Jun 15. PMID 16778145
- [Background] Calado RT, Young NS. Telomere maintenance and human bone marrow failure. Blood. 2008 May 1;111(9):4446-55. doi: 10.1182/blood-2007-08-019729. Epub 2008 Jan 31. PMID 18239083
- [Background] Yamaguchi H, Calado RT, Ly H, Kajigaya S, Baerlocher GM, Chanock SJ, Lansdorp PM, Young NS. Mutations in TERT, the gene for telomerase reverse transcriptase, in aplastic anemia. N Engl J Med. 2005 Apr 7;352(14):1413-24. doi: 10.1056/NEJMoa042980. PMID 15814878
- [Derived] Townsley DM, Dumitriu B, Liu D, Biancotto A, Weinstein B, Chen C, Hardy N, Mihalek AD, Lingala S, Kim YJ, Yao J, Jones E, Gochuico BR, Heller T, Wu CO, Calado RT, Scheinberg P, Young NS. Danazol Treatment for Telomere Diseases. N Engl J Med. 2016 May 19;374(20):1922-31. doi: 10.1056/NEJMoa1515319. PMID 27192671
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-H-0209.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Danazol: Oral administration of Danazol (800 mg daily divided into two doses per day) to be given for 2 years
Period: Overall Study
Arm/Group | Danazol
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Danazol
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 22
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 18
  More than one race | 3
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Having Attenuation of Accelerated Telomere Attrition
Description: The primary efficacy end point was a 20% reduction in the annual rate of telomere attrition measured at 24 months. The biologic response at 24 months, was defined as a reduction in the telomere length attrition rate to 96 bp per year or less. The normal rate of telomere loss of approximately 60 bp per year. Telomere length was determined with a semiautomated, Clinical Laboratory Improvement Amendments (CLIA)-approved real-time quantitative PCR (qPCR) assay performed in triplicate and validated for human cells
Time Frame: 24 months
Population: The analyses included only those subjects who took Danazol
Measure: Count of Participants; unit: Participants
Arm/Group | Danazol
Number analyzed (Participants) | 27
Participants | 12

ADVERSE EVENTS:
Arm/Group | Danazol
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 3/27
Other Adverse Events (participants affected / at risk) | 24/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Danazol (N=27)
Diarrhoea (Gastrointestinal disorders) | 1
Joint swelling (General disorders) | 1
Oedema peripheral (General disorders) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Pneumocystis jirovecii pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Danazol (N=27)
Anaemia (Blood and lymphatic system disorders) | 2
Pallor (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Otitis externa (Ear and labyrinth disorders) | 1
Scleritis (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Decreased appetite (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Infection (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Proctalgia (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 2
Back pain (General disorders) | 1
Cough (General disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 12
Feeling hot (General disorders) | 2
Influenza like illness (General disorders) | 1
Irritability (General disorders) | 1
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Peripheral swelling (General disorders) | 1
Pyrexia (General disorders) | 1
Toothache (General disorders) | 1
Upper respiratory tract infection (General disorders) | 1
Sinus congestion (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Cystitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 2
Tooth disorder (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 2
Viral infection (Infections and infestations) | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Increased tendency to bruise (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1
Umbilical hernia (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 2
Transaminases increased (Investigations) | 1
Weight increased (Investigations) | 4
Iron overload (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Chest discomfort (Musculoskeletal and connective tissue disorders) | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Muscle hypertrophy (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 5
Headache (Nervous system disorders) | 4
Migraine (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 3
Hypersomnia (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Libido increased (Reproductive system and breast disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 4
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 4
Folliculitis (Skin and subcutaneous tissue disorders) | 1
Hirsutism (Skin and subcutaneous tissue disorders) | 1
Hot flush (Skin and subcutaneous tissue disorders) | 1
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Subcutaneous abscess (Skin and subcutaneous tissue disorders) | 1
Haemangioma (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
After 27 patients were enrolled, the study was halted early, because telomere attrition was reduced in all 12 patients who could be evaluated for the primary end point.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes